CLINICAL TRIAL: NCT02741960
Title: A Multicenter, Randomised, Double-blind Placebo Controlled Trial on the Efficacy and Safety of add-on Metformin to Conventional Immunosuppressants in Systemic Lupus Erythematosus
Brief Title: The Effect of Metformin on Reducing Lupus Flares
Acronym: Met Lupus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shuang Ye, Executive Director, Dept. Rheumatology, Renji Hospital South Campus, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHDC12015902
Record Dates: First submitted 2016-04-07; First posted 2016-04-18 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: metformin; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Experimental): Eligible patients for clinical trial were randomized in a 1:1 ratio to metformin/placebo add-on. Subjects randomized to metformin will receive a target dose of 500 mg three times daily. Investigators were allowed to adjust the dose according to the patients' tolerance.
  Interventions: Drug: metformin
- placebo (Placebo Comparator): Eligible patients for clinical trial were randomized in a 1:1 ratio to metformin/placebo add-on. Subjects randomized to placebo will receive a target dose of 500 mg three times daily. Investigators were allowed to adjust the dose according to the patients' tolerance.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: metformin — 500 mg metformin three times daily
  Other Names: Metformin Hydrochloride Tablets
  Arms: metformin
Drug: placebo — 500 mg placebo three times daily
  Arms: placebo

SUMMARY:
This is a multicenter, randomised, double-blind placebo controlled trial on the efficacy and safety of add-on metformin to conventional immunosuppressants in systemic lupus erythematosus (SLE).

The purpose of this study is to evaluate: 1) the effect of metformin on reducing disease flares; 2) the influence of metformin on corticosteroid sparing effect; 3) the influence of metformin on body mass index (BMI); 4) the safety of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Willingness of the subject to participate in the study, proven by signing the informed consent;
* Systemic lupus erythematosus (SLE), as defined by meeting at least 4 of 11 classification criteria of American College of Rheumatology for the classification of systemic lupus erythematosus, either sequentially or coincidentally. The 4 criteria doesn't need to be present at the time of study enrollment;
* The course of SLE longer than1 year; and there is a clear record of disease flares in the past 1 year with prednisone more than 20mg/day;
* Patients with mild/moderate disease activity (score≤ 6 at screening on SLEDAI); no British Isles Lupus Assessment Group (BILAG) A or no more than one B;
* A stable treatment regimen with fixed doses of prednisone (≤ 20mg/day), antimalarial, or immunosuppressive drugs (azathioprine/ mycophenolate mofetil/ methotrexate/ ciclosporin/ leflunomide/ thalidomide) for at least 30 days.

Exclusion Criteria:

* Patients who are unwilling to sign the inform consent;
* Alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) > 2 times upper normal limits; creatinine clearance rate < 60ml/min;
* Patients who used cyclophosphamide 6-months before screening; used biological agents 12-months before screening;
* Previous exposure of metformin within 30 days before screening; or previous history of intolerant to metformin;
* Patients who diagnosed of diabetes mellitus;
* Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
numbers of participants who remained at risk of flares at each visit | one year
  the effect of metformin on reducing disease flares

SECONDARY OUTCOMES:
changes in prednisone dose from baseline at each visit | one year
  the influence of metformin on corticosteroid sparing effect
changes in BMI from baseline at each visit | one year
  the influence of metformin on BMI
number of participants with treatment-related adverse events | one year
  the safety of metformin

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Ye, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Ethics Committee of Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang H, Li T, Chen S, Gu Y, Ye S. Neutrophil Extracellular Trap Mitochondrial DNA and Its Autoantibody in Systemic Lupus Erythematosus and a Proof-of-Concept Trial of Metformin. Arthritis Rheumatol. 2015 Dec;67(12):3190-200. doi: 10.1002/art.39296. PMID 26245802
- [Derived] Sun F, Wang HJ, Liu Z, Geng S, Wang HT, Wang X, Li T, Morel L, Wan W, Lu L, Teng X, Ye S. Safety and efficacy of metformin in systemic lupus erythematosus: a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Rheumatol. 2020 Apr;2(4):e210-e216. doi: 10.1016/S2665-9913(20)30004-7. Epub 2020 Feb 24. PMID 38268156
- [Derived] Sun F, Geng S, Wang H, Wang H, Liu Z, Wang X, Li T, Wan W, Lu L, Teng X, Morel L, Ye S. Effects of metformin on disease flares in patients with systemic lupus erythematosus: post hoc analyses from two randomised trials. Lupus Sci Med. 2020 Oct;7(1):e000429. doi: 10.1136/lupus-2020-000429. PMID 33093216